CLINICAL TRIAL: NCT03534635
Title: An Interventional Phase II Study to Analyze the Modulation of the Tumor Microenvironment by MK-3475 (Pembrolizumab) Using a Systems Biology Approach (PEMSYS)
Brief Title: Analysis of the Modulation of the Tumor Microenvironment by MK-3475 (Pembrolizumab) Using a Systems Biology Approach (PEMSYS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Krisztian Homicsko, MD, PhD, Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-PEMSYS_2017
Record Dates: First submitted 2018-04-19; First posted 2018-05-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Melanoma Naive to Immune Therapy in Metastatic Setting
Keywords: metastatic melanoma; tumor microenvironment; pembrolizumab; PD1
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg will be administered intravenously every 3 weeks, for a maximum of 2 years, until progression, unacceptable toxicity, or withdrawal of consent, whichever happens first.
  Patients may be treated for up to one year of additional treatment with pembrolizumab via the Second Course Phase, and according to defined criteria.
  Interventions: Drug: Pembrolizumab; Drug: Pembrolizumab - additional treatment

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab monotherapy at 200 mg every 3 weeks for 2 years maximum.
  Other Names: anti-PD-1, MK-3475
Drug: Pembrolizumab - additional treatment — Patients may be retreated for one year of additional pembrolizubmab therapy (200 mg every 3 weeks).
  Other Names: anti-PD-1, MK-3475

SUMMARY:
This is a monocentric, prospective, interventional and translational phase II study. Metastatic melanoma (mMEL) patients who are naive to immune therapy in the metastatic setting, and for whom an anti-Programmed Cell Death-1 (PD-1) therapy is needed could be eligible.

The aim of the study is to identify biological markers which allow to better understand and predict the tumor response to pembrolizumab treatment, and thus to establish more efficient treatments for selected patients. Eligible patients will be registered (n=30) and will be treated with pembrolizumab monotherapy at 200 mg every three weeks for 2 years maximum until progression, unacceptable toxicity, or withdrawal of consent, whichever happens first. Patients may be treated for up to one year of additional treatment with pembrolizumab via the Second Course Phase. Patients will be followed medically and radiographically during pembrolizumab treatment. Patients will be followed radiographically every 9 weeks (+/- 7 days) until progression and disease evaluation will be assessed by RECIST 1.1 criteria. After progression, patients will be followed every 6 months for 5 years to collect survival data.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Patients with locally advanced or metastatic treatment naïve incurable metastatic cutaneous melanoma
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion at 3 timepoints (screening, within first 2 months of treatment, and at progression).
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile for the course of the study through at least 4 months after the last dose of study medication.
* Male subjects and their female partners should agree to use 2 methods of contraception starting with the first dose of study therapy through at least 4 months after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Tuberculosis Bacillus), Human Immunodeficiency Virus (HIV); has known active Hepatitis B or Hepatitis C
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.[Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.] [Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.]
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through at least 4 months after the last dose of trial treatment
* Has received prior therapy with an anti-Programmed Cell Death-1 (PD-1), anti-Programmed Cell Death Ligand-1 (PD-L1), or anti-PD-L2 agent in the metastatic setting.
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers using genomics and proteomics tools (single cell RNA analysis, exome sequencing, single cell profiling), multiplexed immunohistochemistry and bioinformatics. | 8 years
  The origin of individual cells of the tumor microenvironment will be identified after single cell analysis at the transcriptional and protein level. Then gene expression from cells derived by tumor biopsies, and from peripheral blood samples, which are collected before and after exposure to MK3475 will be measured, and qualitative and quantitative data will be reported.

SECONDARY OUTCOMES:
Efficacy, in order to define responder and non-responder patients and select translational findings that are associated to clinical outcome. | 8 years
  Secondary outcomes will be derived from analyzes of the primary outcome measures. Tumor response will be evaluated according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided